CLINICAL TRIAL: NCT07131436
Title: The Effect of Equine-Assisted Therapy on Behavior Changes: An Application on Individuals With Autism
Brief Title: Equine-Assisted Therapy in the Behavior of Individuals With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Vesile Şahiner Güler, Principal Investigator, TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ERU-SAGENS-VSG-03
Record Dates: First submitted 2025-07-30; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; autism spectrum disorder; quine-assisted therapy; exercise; behavior; parental opinion
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Motor Activity; Behavior

STUDY DESIGN:
Intervention Model Description: The research was designed in a quantitative study, experimental research method, single group pre-test-post-test, without control group experimental design model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Equine-assisted therapy group (Experimental): The target population of the study consisted of children diagnosed with autism spectrum disorder (ASD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5, 2013) criteria.Autistic children aged 9-11 years with autism spectrum disorder, who were receiving education and rehabilitation services from four private rehabilitation centers in the Güngören, Bayrampaşa, Fatih, and Zeytinburnu districts of Istanbul, were selected from among 184 children diagnosed with autism spectrum disorder. Parents were provided with detailed information about the study and volunteer participants were included in the study. The study group consisted of a total of (n=20) volunteer participants, female (n=10) and male (n=10), with a mean age of 9.90±1.44 years.
  Interventions: Other: Horse therapy

INTERVENTIONS:
Other: Horse therapy — Participating children received horseback riding and riding training twice a week for 30 minutes over an eight-week period. The training included developing body and object use skills, relationship building skills, language skills, social and self-care skills, and sensory skills. These included mounting and dismounting a horse; sitting correctly; holding and using the reins; bustling movements on the horse, forward and backward, sideways, and reaching with the hands; naming printed pictures; reading numbers; throwing objects at targets with the right and left hands; developing a dialogue with the trainer; standing up with and without stepping on the stirrups; sitting down and standing; reaching forward and backward and lying down on the horse; petting the horse with one's hands; trying to touch the horse's front legs with the right and left hands; and holding the horse's mane. At the end of the training, the parents of the participating children completed the Autism Behavior Checklist.

SUMMARY:
Purpose of the Study: The aim of this study was to examine the effects of 8 weeks of equine-assisted therapy exercises applied to children with autism spectrum disorder on autistic behavioral levels (sensory development, relationship building skills, development in body and object use, social and self-care development, and language skills) based on parental opinions.

Materials and Methods: The study group consisted of 20 volunteers (n=20) with a mean age of 9.90±1.44 years. They were diagnosed with ASD according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5, 2013), had partial verbal communication, had not received prior equine-assisted therapy training, had underdeveloped basic life skills (eating and dressing), were not taking regular medication, and had no other chronic diseases other than autism. Participants participated fully in equine-assisted therapy sessions twice a week for 8 weeks.

The study included: Quantitative studies were designed using a single-group pretest-posttest experimental design without a control group, a method used in experimental research methods. A survey was used as the data collection method. Data were collected in three different stages using the Autism Behavior Checklist (ABC) scale, administered face-to-face to the parents of the participating children under the supervision of the researcher. The data were recorded in the SPSS 25 package program. Repeated Measures ANOVA was used as the statistical analysis.

Autism Behavior Checklist (ABC) The Autism Behavior Checklist (ABC) was developed by Krug et al. (1980), and its Turkish adaptation and validity and reliability study were conducted by Irmak et al. (2007). The ABC scale has five factors and 57 items. The scale factors include 9 items on the sensory dimension, 12 items on relationship building, 12 items on body and object use, 13 items on language skills, and 11 items on social and self-care skills. The highest possible score on this scale is 159, and the lowest is 0. In other words, high scores on the scale indicate a high prevalence of autism symptoms. The Autism Behavior Checklist, also known as the ABC, is one of the most frequently used measurement tools for screening and assessing autism (De Bildt et al. 2005). The advantage of the ABC scale in the application process is that it is a scale that makes it possible to obtain information about autistic children from both educators and parents (Krug et al. 1980).Week Day Time Purpose Event Content

1 1 30 min Getting used to the environment and the horses Introduction to the therapy center, observing horses, and practicing getting close to horses 2 30 min First contact with the horse Touching the horse with your hands and holding the horse's mane while watching it 2 1 30 min Basic riding stances Balance exercises by sitting on a horse, learning the correct sitting position 2 30 min Movement awareness Slight bending forward, backward and sideways with the bust

3 1 30 min Upper body and arm coordination Extending the hands forward, to the sides and to the feet, petting the horse 2 30 min Lying on a horse Lying forward and backward, on the back or face down 4 1 30 min Motor skills Attempts to stand up with or without stepping on the stirrups 2 30 min Object control Games of throwing objects at targets with the right/left hand 5 1 30 min Social interaction Communicating with the coach (greeting, saying your name) 2 30 min Sensory awareness Touching the horse's front legs, noticing the mane, hugging the horse 6 1 30 min Balance and direction Trials of turning left and right, forward and backward, and steering on a horse 2 30 min Audiovisual mapping Saying the names of printed images and number recognition exercises 7 1 30 min Integration of mixed skills Trials of rein holding, steering and basic commanding 2 30 min Mixed-task applications Multitasking involving throwing objects + talking + changing direction 8 1 30 min Skill reinforcement Integrated repetition of all learned movements 2 30 min Skill reinforcement Integrated repetition of all learned movements 10 - - Final observation and evaluation Completing the Parent Autism Behavior Checklist Scale

DETAILED DESCRIPTION:
Equine-assisted therapy training for individuals with autism is not a standalone method. It is part of a treatment and education program that aims to address the individual's physical, mental, emotional, and spiritual well-being as a whole. In addition to the sensory and motor benefits of being on a horse, basic sports skills practiced on horseback (such as throwing and catching a ball, ring spinning, gross motor imitation skills, hand-eye coordination, directional training, etc.) will also provide physical and physiological benefits to individuals with disabilities. Autism is defined as a neurodevelopmental disorder that develops at birth or in the early years of life, manifesting itself as a lack of social skills, repetitive behaviors, difficulties with verbal and nonverbal communication, and motor performance deficits. The problems and effects observed in individuals with autism vary according to age and developmental level. Limited motor coordination, fine and gross motor function deficits, repetitive movements, auditory and visual hypersensitivity or decreased auditory and visual sensitivity, inability to maintain postural orientation, inability to plan movement, and inability to integrate sensory stimuli are observed in individuals of different ages and developmental levels. At the same time, sensory and perceptual problems and different cognitive developments lead to repetitive, stereotypical, and restricted body movements. Individuals with autism spectrum disorder exhibit deficits in postural control, gait, upper and lower extremity coordination, and fine motor skills. These deficits can lead to difficulties with verbal commands and tool use.The target population for the study consisted of children diagnosed with autism spectrum disorder (ASD) according to the Diagnostic and Statistical Manual of Mental Disorders criteria. For the purpose of the study, homogeneous sampling, a purposive sampling method, was used to include individuals with similar characteristics in the sample. The homogeneous sampling method is used to identify a distinct subgroup by creating a small, similar sample.Training process and post-test phase: Before starting the training, the participating children and their parents were introduced to the therapy center and observed the therapy horses to help them adapt. The participating children received horseback riding and riding training twice a week for 30 minutes over an eight-week period. The training included body and object use skills, relationship building skills, language skills, social and self-care skills, and developing sensory skills, including mounting and dismounting a horse; sitting correctly; holding and using the reins; bustling movements on the horse, forward and backward, sideways, and reaching with the hands; naming printed pictures; reading numbers; throwing objects at targets with the right and left hands; developing dialogue with the trainer; standing up with and without stepping on the stirrups; sitting down and standing; reaching forward and backward and lying down on the horse; petting the horse with one's hands; trying to touch the horse's front legs with the right and left hands; and holding the horse's mane. At the end of the training, the parents of the participating children completed the Autism Behavior Checklist (ABC) under the researcher's supervision. The training sessions were conducted considering the age, gender, and housing status of the autistic children.Research data were collected in three stages. In the first stage, parents of autistic children were provided with detailed information about the study and administered a pre-test of the Autism Behavior Checklist Scale. The pre-test included parents rating their children's behavior before receiving the training. In the second stage, the autistic children were taught how to mount and dismount, sit correctly, hold and use the reins, move left and right and forward and backward while riding, reach forward and backward with their hands, sideways and feet, name printed pictures, read numbers, throw objects with their right and left hands to target targets, develop a dialogue with their trainer, stand up with and without stirrups, sit down and stand up, lie down and lie down on the horse, pet the horse with their hands, try to touch the horse's front legs with their right and left hands, and hold the horse's mane. The post-test included parents rating their children's behavior after receiving the training. In the third stage, children with autism who completed their equine-assisted therapy training continued their normal life and education for two weeks and were observed by their parents. In the tenth week, the Autism Behavior Checklist Scale permanence test measurements were applied to the parents under the supervision of the researcher and the research data collection process was completed.Application of Data Collection Instruments (Experimental Procedure) Participating children received 480 hours of training over an eight-week period, twice a week, for 16 sessions. Each session lasted 30 minutes. The therapy training for children with autism was conducted individually and was conducted by a psychologist, a physiotherapist, a horse trainer, and two walker personnel.

The data collection process consisted of three phases.

1. Pretest Phase: In this phase, the parents of the children included in the study were informed about the tests to be conducted and had them complete the Autism Behavior Checklist (ABC) under the supervision of the researcher and with the parents' active participation.
2. Training Process and Posttest Phase: Before the training began, the participating children and their parents were interviewed and observed therapy horses to familiarize themselves with the therapy center and to help them adapt to the center. Participating children received horseback riding and riding training twice a week, lasting 30 minutes, for an eight-week period. The training included body and object use skills, relationship building skills, language skills, social and self-care skills, and developing sensory skills, including mounting and dismounting a horse; sitting correctly; holding and using the reins; bustling movements on the horse, forward-backward, side-to-side, and reaching movements with the hands; naming printed images shown to the child; reading numbers; throwing objects to targets with the right and left hands; developing dialogue with the trainer; standing up with and without stepping on the stirrups; sitting down and standing; reaching forward and backward and lying down on the horse; petting the horse with one's hands; trying to touch the horse's front legs with the right and left hands; and holding the horse's mane. At the end of the training, the parents of the participating children completed the Autism Behavior Checklist (ABC) scale under the supervision of the researcher. The training was conducted considering the age, gender, and housing status of the autistic children. 3- Testing the permanence of the effect: Children who completed the therapy training were observed by their parents starting from the week the training ended, and after two weeks (in the 10th week), a permanence test was conducted by having the parents fill out the autism behavior checklist (ABC) scale again under the supervision of the researcher.Autism Behavior Checklist (ABC) The Autism Behavior Checklist (ABC) was developed by Krug et al. and its Turkish adaptation and validity and reliability study were conducted by Irmak et al. The ABC scale has five factors and 57 items. The scale factors include 9 items on the sensory dimension, 12 items on relationship building, 12 items on body and object use, 13 items on language skills, and 11 items on social and self-care skills. The highest possible score on this scale is 159, and the lowest is 0. In other words, high scores on the scale indicate a high prevalence of autism symptoms. The Autism Behavior Checklist, also known as the ABC, is one of the most frequently used measurement tools for screening and assessing autismThe advantage of the Autism Behavior Checklist Scale in the application process is that it is a scale that makes it possible to obtain information about autistic children from both educators and parents.

Statistical Analysis Data obtained from the Autism Behavior Checklist (ABC) scale pre-, post-, and retention test measurements were transferred to the IBMM SPSS 25 program. The normal distribution curves of the scores, skewness-kurtosis values, and the Shapiro-Wilk test values used when the group size was less than 30 were examined using histograms obtained from the scale. The data were determined to be normally distributed. The "Repeated Measures Anova" test statistic, used for repeated measurements, was applied to reveal the significance between the Autism Behavior Checklist (ABC) scale pre-test, post-test, and retention test values based on parental opinions. The sphericity assumption was implemented using the Mauchly test, and the "Sphericity Assumed" test values were taken into account. Furthermore, the "Benferroni" test statistic was used in pairwise comparisons to determine between which measurements the statistical difference occurred. The calculation (d) value developed by Cohen was used to interpret the calculated effect size. If the (d) value is less than 0.2, the effect size can be defined as weak; if the (d) value is 0.5, the effect size can be defined as medium; and if the (d) value is greater than 0.8, the effect size can be defined as strong.

ELIGIBILITY:
Inclusion Criteria:

1. Having been diagnosed with ASD according to DSM-5 criteria,
2. Having partial verbal communication,
3. Not having received previous equine-assisted therapy training,
4. Not having developed basic life skills (eating and dressing),
5. Not taking regular medication,
6. Not having any other chronic disease other than autism.

Exclusion Criteria:

1. Having a chronic disease other than autism,
2. Not attending therapy training twice in a row,
3. Weighing more than 60 kg during the training period.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Autism Behavior Checklist (ABC) | 10-week period with therapy applied for 8 weeks and parents' opinions on the permanence effect obtained 2 weeks later.
  The Autism Behavior Checklist (ABC) was developed by Krug et al. (1980), and its Turkish adaptation, validity, and reliability studies were conducted by Irmak et al. (2007). The ABC scale has five factors and 57 items. The scale factors include 9 items for the sensory dimension, 12 items for establishing relationships, 12 items for body and object use, 13 items for language skills, and 11 items for social and self-care skills. The highest score possible on this scale is 159, and the lowest is 0. In other words, high scores on the scale indicate a high prevalence of autism symptoms. The Autism Behavior Checklist, an autism behavior checklist, is one of the most frequently used measurement tools for screening and assessing autism and is referred to as the ABC (De Bildt et al. 2005). The advantage of the ABC scale in the application process is that it is a scale that makes it possible to obtain information about autistic children from both educators and parents (Krug et al. 1980).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Behzat Turan, Associate Professor, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Talas, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the data collected from children.